CLINICAL TRIAL: NCT06949449
Title: Upper Limb Functional Capacity in Individuals Diagnosed With Mental Disorders: A Cross-Sectional Study
Brief Title: Upper Limb Function in Mental Health Disorders
Acronym: UFMC-MH2025
Status: Completed | Type: Observational
Sponsor: Universidad de Burgos (Other)
Responsible Party: Sponsor
Other Study IDs: UFMC-MH2025; IO 50/2024 (Other: Universidad de Burgos)
Record Dates: First submitted 2025-04-08; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-11

CONDITIONS: Mental Health; Multiple Sclerosis
Keywords: mental disorders; upper extremity; hand strength; motor skills; hand
MeSH Terms: conditions — Psychological Well-Being; Multiple Sclerosis; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- EXPERIMENTAL GROUP: Participants diagnosed with a mental disorder (MD). Evaluated for upper limb functionality, including strength, fine and gross manual dexterity, sensitivity, tactile discrimination, and performance in activities of daily living (ADL).
- CONTROL GROUP: Participants without any diagnosed mental disorder. Assessed using the same measures to serve as a baseline for comparison with the MD group.

SUMMARY:
Background: Individuals with mental disorders (MD) often experience motor issues, yet upper limb functionality remains understudied.

Objective: To compare upper limb function in individuals with and without MD, focusing on motor capacity, dexterity, and performance.

Design: Cross-sectional, qualitative, multicenter study. Methods: Assessed strength, motor skills, sensitivity, and daily function. Used T-test, Mann-Whitney U, Spearman correlation, and Chi-square.

DETAILED DESCRIPTION:
Background: Research suggests individuals with mental disorders (MD) often face motor difficulties, such as issues with gait and posture. However, there is limited research on upper limb functionality in the mental health context.

Objective: To compare upper limb functionality between individuals with and without MD, focusing on differences in motor capacity, manual dexterity, and functional performance.

Study Design: Cross-sectional, qualitative, multicenter study.

Methods: Strength, fine and gross motor skills, sensitivity, tactile discrimination, and were assessed, along with functional limitations in daily activities. Statistical methods used included independent samples T-test, Mann-Whitney U test, Spearman correlation, and Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

Mental Disorder Group

* Participants with a mental disorder (MD) had to meet the following criteria:
* A formal diagnosis of a mental disorder according to the DSM-V.
* Aged between 18 and 65 years.
* Treatment stability, defined as being under stable pharmacological and psychiatric treatment for at least three months.
* Clinical stability, meaning no acute psychiatric episodes in the last three months that could interfere with participation in the study.
* Ability to follow instructions and communicate effectively, confirmed by scoring at least 23 points on the Mini-Mental State Examination (MMSE).

Control Group (Healthy Participants)

* Healthy individuals were required to meet the following inclusion criteria:
* Aged between 18 and 65 years.
* Ability to follow instructions and communicate effectively, also defined by a minimum MMSE score of 23.

Exclusion Criteria:

* Presence of neurological conditions, such as multiple sclerosis, stroke, or similar disorders.
* History of upper limb rehabilitation within the past six months.
* Any acute or chronic condition affecting the upper limb that could interfere with the results, including but not limited to arthritis, osteoarthritis, or carpal tunnel syndrome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of 38 participants was obtained, consisting of 19 individuals diagnosed with a mental disorder (MD) and 19 healthy controls.
  Initially, 40 participants were contacted; however, two were unable to participate due to scheduling conflicts that prevented them from completing the assessment.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Nine Hole Peg Test (NHPT) | 3 weeks
  Assesses fine manual dexterity. Participants place and remove nine pegs from holes as quickly as possible, using one hand at a time. The test is performed twice, and the average time is recorded. Lower scores indicate better fine motor skills.
  The NHPT has shown high test-retest reliability, inter-rater reliability, and internal consistency in previous studies, including Spanish-speaking populations.
Box and Block Test (BBT) | 3 weeks
  Measures gross manual dexterity. Participants move as many blocks as possible from one compartment of a box to another in one minute, using each hand separately. Blocks must be moved over a dividing wall without throwing or bumping. Higher scores indicate better gross dexterity.
  The BBT is widely used and validated across different populations.
Digital Hand Dynamometer | 3 weeks
  Evaluates grip strength. Participants squeeze a hydraulic hand dynamometer three times with each hand while seated with the elbow at 90°. The average of the three trials is used. Higher scores indicate greater grip strength.
  This test has strong validity, sensitivity, and reliability, including among Spanish-speaking populations.
Semmes-Weinstein Monofilament Test | 3 weeks
  Assesses tactile sensitivity. Monofilaments of varying thickness are applied to specific areas of the hand (fingertips, palm, back of the hand). The finest filament perceived consistently (at least 2 out of 3 times) is recorded as the sensitivity threshold.
  There is limited psychometric data available in Spanish-speaking populations, though the test is widely used clinically.
Two-Point Discrimination Test (Touch-Test) | 3 weeks
  Evaluates tactile discrimination ability. Two points are applied to the skin at decreasing distances until the participant can no longer distinguish them as separate. Tested on the same hand areas as the monofilament test.
  It assesses the density of tactile receptors and sensory pathway integrity. Psychometric properties in Spanish-speaking populations are not well established.
QuickDASH Questionnaire | 3 weeks
  A shortened version of the DASH questionnaire, designed to evaluate disability and symptoms in the upper limb. It consists of 11 items rated on a 5-point scale. Higher scores indicate worse functional ability.
  Both the original and Spanish versions have demonstrated good reliability, internal consistency, sensitivity to change, and construct validity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Burgos, Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) that underlie the results reported in this study-including anonymized data on motor assessments, functional performance, and demographic variables-will be made available upon reasonable request to qualified researchers.
  Requests include a clear research purpose and it is reviewed and approved by the principal investigator and the ethics committee, ensuring data privacy and compliance with relevant regulations. Data will be shared in a de-identified format to protect participant confidentiality.
Supporting Information: Study Protocol, ICF
Time Frame: The IPD will be made available upon reasonable request to qualified researchers.
  Start date for data availability: January 1, 2026
  End date for data availability: December 31, 2030
Access Criteria: Qualified researchers affiliated with academic institutions, healthcare organizations, or research centers will be eligible to request access to the individual participant data (IPD) and supporting documentation. Access will be granted for non-commercial, scientific research purposes only.
URL: https://www.ubu.es/tecnologia-y-terapia-ocupacional-tecto-0

REFERENCES:
- [Background] Jiang R, Westwater ML, Noble S, Rosenblatt M, Dai W, Qi S, Sui J, Calhoun VD, Scheinost D. Associations between grip strength, brain structure, and mental health in > 40,000 participants from the UK Biobank. BMC Med. 2022 Sep 9;20(1):286. doi: 10.1186/s12916-022-02490-2. PMID 36076200
- [Background] Desrosiers J, Bravo G, Hebert R, Dutil E, Mercier L. Validation of the Box and Block Test as a measure of dexterity of elderly people: reliability, validity, and norms studies. Arch Phys Med Rehabil. 1994 Jul;75(7):751-5. PMID 8024419
- [Background] Moreno-Morente G, Hurtado-Pomares M, Sanchez-Perez A, Terol-Cantero MC. Translation, Cross-Cultural Adaptation, and Feasibility of the NHPT-E of Manual Dexterity for the Spanish Population. Healthcare (Basel). 2024 Feb 27;12(5):550. doi: 10.3390/healthcare12050550. PMID 38470661
- [Background] Walther S, Mittal VA, Stegmayer K, Bohlhalter S. Gesture deficits and apraxia in schizophrenia. Cortex. 2020 Dec;133:65-75. doi: 10.1016/j.cortex.2020.09.017. Epub 2020 Oct 3. PMID 33099076
- [Background] Vale N, Gandolfi M, Mazzoleni S, Battini E, Dimitrova EK, Gajofatto A, Ferraro F, Castelli M, Camin M, Filippetti M, De Paoli C, Picelli A, Corradi J, Chemello E, Waldner A, Saltuari L, Smania N. Characterization of Upper Limb Impairments at Body Function, Activity, and Participation in Persons With Multiple Sclerosis by Behavioral and EMG Assessment: A Cross-Sectional Study. Front Neurol. 2020 Feb 14;10:1395. doi: 10.3389/fneur.2019.01395. eCollection 2019. PMID 32116983